CLINICAL TRIAL: NCT06991413
Title: Pilot Study to Investigate the Impact of an App on the Quality of Life and Symptoms of Individuals Affected by Premenstrual Syndrome
Brief Title: Impact of an App on the Quality of Life and Symptoms in Individuals With Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endo Health GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RCT_PilotPMS
Record Dates: First submitted 2025-04-28; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-04

CONDITIONS: Premenstrual Syndrome; Premenstrual Syndrome-PMS
Keywords: Digital Therapeutics; Premenstrual syndrome (PMS)
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care-as-usual (No Intervention): Control group has access to care-as-usual only
- Care-as-usual + digital PMS app (Experimental): The intervention group has access to the PMS app and its functions in in addition to care-as-usual
  Interventions: Device: PMS App

INTERVENTIONS:
Device: PMS App — The PMS App helps to implement multimodal self help measures in the daily lives of PMS patients through various functions such as symptom diary and interactive exercises.
  Arms: Care-as-usual + digital PMS app

SUMMARY:
This pilot study explored the effectiveness and acceptance of a digital app for the self-management of PMS. A total of 175 participants were randomized into an intervention and a control group. Findings indicate that the app offers beneficial effects on PMS-specific symptoms and broader health aspects such as fatigue and emotional well-being. The study also provided valuable insights for the design of future larger trials and highlights the promising potential of the app to enhance individualized care.

ELIGIBILITY:
Inclusion Criteria:

* Legal capacity
* Residency in Germany
* Female gender
* Age ≥18 years
* Diagnosed and medically confirmed current PMS (N94.3)
* Ownership of a smartphone and ability to use it
* Internet access for app usage and questionnaire completion
* Email address for registration
* Willingness to complete questionnaires online
* Motivation for regular app usage
* Sufficient proficiency in the German language

Exclusion Criteria:

* Pregnancy, breastfeeding, or the onset of menopause during the study period
* Changes in hormonal therapy and/or use of antidepressants within eight weeks prior to the study start and/or planned in the upcoming 12 weeks
* Previous or current access to the Endo-App or other comparable digital health applications, or current active prescription
* Current participation in other clinical studies
* Failure to meet the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
PMS-Impact Questionnaire (PMS-I) | 12 weeks
  PMS-specific impairments, min = 18 and max=72, higher scores indicate a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Endo Health GmbH, Chemnitz, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No